CLINICAL TRIAL: NCT02232256
Title: A Phase 3 Double Blind, Randomized, Placebo Controlled, Cross-Over Trial to Asses the Efficacy of CALPXT96™in Improving Sleep Quality in Patients With Chronic Non-cancer Pain
Brief Title: The Efficacy of CALPXT96™in Improving Sleep Quality in Patients With Chronic Non-cancer Pain
Acronym: CALPXT96
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Site unable to enrol recruited subjects
Sponsor: 9305-9954 Quebec Inc (Industry)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CALPXT96-01
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain; Insomnia
Keywords: Chronic non-cancer pain; Insomnia; California poppy; Eschscholzia californica; Pain; Sleep quality
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CALPXT96 (Experimental): 1. 1st treatment period: 4 weeks CALPXT96 (two capsules hs at bedtime)
  2. 2 week wash out period
  3. 2nd treatment period: 4 weeks placebo (two capsules hs at bedtime)
  Interventions: Drug: CALPXT96
- Placebo (Placebo Comparator): 1. 1st treatment period: 4 weeks placebo (two capsules hs at bedtime)
  2. 2 week wash 'out' period
  3. 2nd treatment period: 4 weeks CALPXT96 (two capsules hs at bedtime)
  Interventions: Drug: CALPXT96

INTERVENTIONS:
Drug: CALPXT96 — Arm 1: intervention begins with CALPXT96 Arm 2: intervention begins with placebo
  Other Names: California poppy standardized extract

SUMMARY:
California Poppy has been traditionally used in Herbal Medicine as an analgesic, mild sedative and/or sleep aid. However there are no human clinical trial data to support its use. Sleep disturbances are a well-recognized component of chronic pain, and lead to additional social withdrawal, greater pain and worsening depression. Most hypnotics available either place the patient at further risk (e.g. benzodiazepines combined with opioids increase the risk of central or obstructive sleep apnea), increase adverse events (dry mouth, daytime somnolence, etc.) or induce sleep but do not improve the quality of sleep (no increase in Rapid Eye Movement or curative sleep). This study intends to use California Poppy to avoid adverse effects while improving sleep. An open-label clinical trial was performed to obtain preliminary safety and efficacy information of California poppy. This trial was approved by a central ethics review board. The study results showed that California poppy, can be used as a co-analgesic to provide additional analgesia and/or sleep improvement to the patient. Patients who are referred to the clinic will be asked to complete a few short questionnaires at every visit and on monthly basis respectively. This data, in addition to the usual follow-up questionnaires used by the clinics' physicians (McGill Pain Intensity, Pain Disability Index, Short-form Health Survey-12v2) and general demographic and medical information will be used to assess California Poppy's effectiveness on patients

DETAILED DESCRIPTION:
Study Design:

This will be an 'n of 1' model, with the patient acting as their own control. To identify any possible negative 'wash out' effect after cessation of the active medication (that could negatively impact the 'no drug' arm) we have to do the following. After baseline documentation with standardized scales, randomize to one of 2 arms:

1. Arm A

   * 1st treatment period: 4 weeks active drug (two capsules of CALPXT96 hs)
   * 2 week wash out period
   * 2nd treatment period: 4 weeks placebo (two capsules of CALPXT96 hs)
2. Arm B

   * 1st treatment period: 4 weeks placebo (two capsules of CALPXT96 hs)
   * 2 week ash out period
   * -2nd treatment period: 4 weeks active drug (two capsules of CALPXT96 hs)

Objectives:

Primary objective

The primary objective of this study is:

* Does nightly use of CALPXT96 improve sleep in patients with CNCP? Secondary objective
* The secondary objective of this study are:
* Does CALPXT96 improve functionality as defined by the PDI (or Short-Form Health Survey-12 (SF12))?
* Does CALPXT96 decrease pain levels (average, highest, lowest) (Brief Pain Inventory)?
* Does CALPXT96 allow for a decrease in other medications prescribed for pain?

Efficacy Measures

* Changes in quality of seep as measured by the the Pittsburgh Sleep Quality Index (PSQI) and the Pain and Sleep Questionnaire (PSQ-3).
* Changes in pain intensity scores (Brief Pain Inventory) and changes in functionality and health related quality of life as measured with the Pain Disability Index (PDI) and SF-12v2 respectively.

Population:

Chronic pain patients suffering from CNCP for greater than 1 year, with complaint of poor sleep (defined as >/= 5 on the Pittsburgh Sleep Quality Index (PSQI), aged 18 and up and of a normal mix of gender, age, and socioeconomic status and with a stable pain management treatment for at least one month.

Inclusion Criteria

Subjects are eligible to be included in the study only if they meet all of the following criteria:

1. Age > 17 and < 75
2. Chronic non-cancer pain (CNCP) associated with a complaint of poor sleep. (Validated tool the Pittsburgh Sleep Quality Index (PSQI) for sleep dysfunction and using a suitable cut points (PSQI >/=5) to ensure greater homogeneity of the sample and the recruitment of only those with significant pain related sleep disturbance.)
3. Stable pain management therapy for 1 month prior to entry into the study
4. Having a confirmed diagnosis of CNCP for greater than 1 year
5. Written informed consent obtained.
6. Subject agreed to follow the protocol.

Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

1. Taking a hypnotic medication at time of enrollment. Patients may be enrolled if they are willing to cease any current hypnotic for at least 2 weeks prior to commencing the study
2. Current alcohol abuse or other addiction
3. Sleep apnea disorder
4. Inability to understand and comply with the instructions of the study
5. Previous enrollment in the study
6. Renal and/or liver insufficiency
7. Patients less than age 18
8. Pregnancy or lactation
9. Current (</=one year) Diagnostic and Statistical Manual-IV (DSM-IV) Axis I diagnosis of major depressive disorder, dysthymia, generalized anxiety disorder and DSM-IV diagnosis of mania, bipolar disorder, or psychosis determined either by patient history

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 and < 75
* Chronic non-cancer pain (CNCP) associated with a complaint of poor sleep. Validated tool the Pittsburgh Sleep Quality Index (PSQI) for sleep dysfunction and using a suitable cut points (PSQI >/=5) to ensure greater homogeneity of the sample and the recruitment of only those with significant pain related sleep disturbance.
* Stable pain management therapy for 1 month prior to entry into the study
* Having a confirmed diagnosis of CNCP for greater than 1 year
* Written informed consent obtained.
* Subject agreed to follow the protocol.

Exclusion Criteria:

* Taking a hypnotic medication at time of enrollment. Patients may be enrolled if they are willing to cease any current hypnotic for at least 2 weeks prior to commencing the study
* Current alcohol abuse or other addiction
* Sleep apnea disorder
* Inability to understand and comply with the instructions of the study
* Previous enrollment in the study
* Renal and/or liver insufficiency
* Patients less than age 18
* Pregnancy or lactation
* Current (</=one year) DSM-IV Axis I diagnosis of major depressive disorder, dysthymia, generalized anxiety disorder and DSM-IV diagnosis of mania, bipolar disorder, or psychosis determined either by patient history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Does nightly use of CALPXT96 improve sleep in patients with CNCP? | Change from Baseline in PSQI at Days 30, 44 and 74.
  Changes in quality of sleep as measured by the the Pittsburgh Sleep Quality Index (PSQI).
Does nightly use of CALPXT96 improve sleep in patients with CNCP? | Change from Baseline in PSQ-3 at Days 15, 30, 44, 59 and 74.
  Changes in quality of sleep as measured by the Pain and Sleep Questionnaire (PSQ-3).

SECONDARY OUTCOMES:
Does CALPXT96 improve functionality as defined by the PDI (or SF12)? | Change from Baseline in PDI (or SF12) at Days 15, 30, 44, 59 and 74.
  Changes in functionality and health related quality of life as measured with the Pain Disability Index (or SF-12v2).
Does CALPXT96 decrease pain levels (average, highest, lowest) (Brief Pain Inventory)? | Change from Baseline in BPI at Days 15, 30, 44, 59 and 74.
  Changes in pain intensity scores (Brief Pain Inventory).
Does CALPXT96 allow for a decrease in other medications prescribed for pain? | Change from Baseline at Days 15, 30, 44, 59 and 74.
  Concomitant and rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: James Ducharme, MD CM, Principal Investigator — McMaster University
Locations (1):
- CPM - Centres for Pain Managemen, Mississauga, Ontario, Canada